CLINICAL TRIAL: NCT01650870
Title: A Single Center, Randomized, Single-blind Pilot Study to Determine the Safety, Efficacy, and Patient Preference of Split-Dose Regimen of Crystalline Lactulose for Cleansing of the Colon as a Preparation for Colonoscopy in Adults
Brief Title: Safety, Efficacy, and Patient Preference of Split-Dose Crystalline Lactulose as a Preparation for Colonoscopy in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other); Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SplitDose Cryst. Lactulose
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Colonoscopy
Keywords: Cathartics; Laxatives; Lactulose; Gastrointestinal Agents; Therapeutic Uses; Pharmacologic Actions

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Evening Only (full-dose) (Active Comparator): The dosing regimen of Crystalline lactulose will be four 45-gram doses (one dose every 60 minutes for 4 straight hours) taken the evening before the colonoscopy procedure.
  Interventions: Drug: Crystalline Lactulose
- Split-dose (Experimental): The dosing regimen of Crystalline lactulose will be three 45-gram doses (one dose every 60 minutes for 3 straight hours) taken the evening before the colonoscopy procedure followed by one 45-gram dose the morning before the colonoscopy procedure.
  Interventions: Drug: Crystalline Lactulose

INTERVENTIONS:
Drug: Crystalline Lactulose

SUMMARY:
The purpose of this study is to determine the efficacy of a split-dose regimen of crystalline lactulose for cleansing of the colon as a preparation for colonoscopy, as assessed by the physician's determination of the cleanliness of the colon using the Boston Bowel Prep Scale (BBPS).

DETAILED DESCRIPTION:
This is a single center, open-label, pilot study to determine the safety, efficacy, and patient preference of a split-dose regimen of Crystalline Lactulose for cleansing of the colon prior to colonoscopy. Safety will be assessed by the occurrence of any treatment emergent adverse events. Efficacy will be determined by the endoscopist's rating of the cleanliness of the colon and the incidence of treatment failure (insufficient evacuation of the bowel). Patient preference will be determined by the patient's responses on a patient questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring bowel evacuation for colonoscopy

Exclusion Criteria:

* Patients with galactosemia (galactose-sensitive diet)
* Patients known to be hypersensitive to any of the components of Crystalline Lactulose
* Patients with a history of a failed bowel preparation
* Patients with severe constipation, defined as those patients taking daily prescription or over-the-counter laxatives
* Patients with possible bowel obstruction, previous colonic surgery, gastric retention, bowel perforation, toxic colitis, toxic megacolon, or ileus
* Patients on lactulose therapy or receiving any treatment for chronic constipation
* Patients less than 18 years of age
* Inability to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]) and agree to abide by the study restrictions
* Be pregnant or nursing
* Be otherwise unsuitable for the study, in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Cleanliness of the Colon During Colonoscopy | Day of the procedure
  To evaluate the primary objective of efficacy of the split-dose, the following endpoint will be measured:
  o Physician's determination of the cleanliness of the colon will be evaluated by completion of the Boston bowel prep scale.

SECONDARY OUTCOMES:
Treatment Failures | Day of the procedure
  To evaluate the secondary objective of efficacy, the following endpoint will be measured:
  o The number and percentage of patient's who by the physician's determination are considered treatment failures (patients with insufficient evacuation of the bowel=Boston bowel prep score < 5, and/or any colon segment score of 0).
Patient Tolerability and Preference | Day before and day of colonoscopy
  To evaluate the secondary objective of patient tolerability and preference on the basis of the following assessments: Patient tolerability and preference questionnaire including 100 mm Visual Analog Scale (VAS) and Likert Scale
Colonic Hydrogen and Methane Gas Production | Day of colonoscopy
  To evaluate the secondary objective of measuring colonic hydrogen and methane gas production as measured by:
  o Colonic hydrogen and methane gas levels.
Safety/Adverse Events | Day before colonoscopy till 7 days after colonoscopy
  To evaluate the secondary objective of safety as measured by the incidence of treatment emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Otto Lin, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical Center, Seattle, Washington, United States